CLINICAL TRIAL: NCT05736809
Title: Comparative Effects of Calcaneal Low Dye Taping Plantar Fascial Stretching and Sham Taping on Acute Plantar Heal Pain and Functional Activity Level in Football Players
Brief Title: Calcaneal Low Dye Taping Plantar Fascial Stretching and Sham Taping in Football Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 30162
Record Dates: First submitted 2023-01-04; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Sports Physical Therapy
Keywords: Calcaneal Taping, ,; Plantar Fascia,; Low Dye Taping; Foot,

STUDY DESIGN:
Intervention Model Description: The study would be a RCT (Randomized control trial) at Pakistan sports board in which convenience sampling technique would be used .This study include total 21 participants and for this purpose lotare method would be used to select the participants on comparison of calcaneal taping , planter fascia stretching and sham taping for one week for acute treatment . Each groups contain 7 participants with heel pain with baseline treatment will be given to each of the groups .
Masking Description: Planter fascia is a fibrous connective tissue originate from the medial calcaneal tubercle and help support the arch of the foot repetitive tensile overload from standing for long periods of time or running causes changes in the aponeurosis. Patient mostly present with pain on first step in the morning or after long non-weight bearing, Tenderness to anterior medial head. Its can first be treated conservatively where 90 % cases treated greater then 6 months of duration. Baseline treatment is given as Rest , Ice , compression and Elevation , with this NSAID ,shoe inset ,Taping, orthotics, deep friction massage and precautions are advised to the patients. Arch taping is most probably used and orthotics in acute treatment is commonly preferred due to its cost.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-Dye taping (Experimental): out of 21 participants 7 will be included in the study design as an experimental group using low-dye taping in acute stage
  Interventions: Other: Low-dye taping
- Plantar fascia stretching (Active Comparator): out of 21 participants 7 will be included in the study design as an active participants group using plantar fscia stretching in acute stage
  Interventions: Other: Plantar fascia stretching
- Sham taping (Placebo Comparator): out of 21 participants 7 will be included in the study design as an active participants group using plantar fscia stretching in acute stage
  Interventions: Other: sham taping

INTERVENTIONS:
Other: Low-dye taping — Low-dye taing using 4 tapes around calcaneam
  Arms: Low-Dye taping
Other: Plantar fascia stretching — out of 21 participants 7 will be included in the study design as an active participants group using plantar fscia stretching in acute stage
  Arms: Plantar fascia stretching
Other: sham taping — out of 21 participants 7 will be included in the study design as an plecebo group using sham taping in acute stage
  Arms: Sham taping

SUMMARY:
Showing the effect of calcaneal Low-dye Taping on acute planter heel pain and functional activity level in football players.

DETAILED DESCRIPTION:
Planter fascia is a fibrous connective tissue originate from the medial calcaneal tubercle and help support the arch of the foot repetitive tensile overload from standing for long periods of time or running causes changes in the aponeurosis. Patient mostly present with pain on first step in the morning or after long non-weight bearing , Tenderness to anterior medial head. Its can first be treated conservatively where 90 % cases treated greater then 6 months of duration. Baseline treatment is given as Rest , Ice , compression and Elevation , with this NSAID ,shoe inset ,Taping, orthotics, deep friction massage and precautions are advised to the patients. Arch taping is most probably used and orthotics in acute treatment is commonly preferred due to its cost.Taping effects most probably overlooked in general gait parameters, patient feedback on pain relief and function recovery.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female football players
* Age (20-45 yrs)
* Pain with the first step upon walking
* Pain located at the heel or Planter surface of Mid-foot consistent with Planter fasciitis
* Presence of an everted calcaneus greater than or equal to 2°

Exclusion Criteria:

* Patient with surgery and treatment with previous 6 month
* History of Ankle or foot fracture
* Congenital deformity of the foot and ankle
* Sever Spasticity
* Use of an Assistive device
* Bilateral Planter heel pain
* Refusal to participate in study

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
numeric pain rating scale | 3 week
  The Numeric Pain Rating Scale (NPRS) is a famous strategy to evaluate Pain. The NPRS has a dependable, substantial and delicate instrument to survey torment. Torment score as per the NPRS (0-10), made during the principal strides toward the beginning of the day, was the essential result (0 as "no aggravation" and 10 as "exceptionally serious agony").
foot and ankle disability index | 3 week
  It is utilized to evaluate the utilitarian restrictions connected with foot and lower leg, action of day to day living and most troublesome errand that are vital for sports e.g., Walk, word related execution, Agony, Rest and Strength. The foot and ankle disability index (FADI) is scored out of 104, with a score of 0 indicating maximum disability and a score of 104 indicating no disability. The total FADI score corresponds to the sum of Activity and Pain subscale scores (maximum score of 88 for Activity and 16 for Pain).

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Dr Tariq, Phd, Principal Investigator — Riphah International University
Locations (1):
- Surya Azeem Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No